CLINICAL TRIAL: NCT02119702
Title: Adolescent Master Protocol for Participants 18 Years of Age and Older (AMP Up)
Acronym: AMP Up
Status: Completed | Type: Observational
Sponsor: Harvard School of Public Health (HSPH) (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH); National Institute on Drug Abuse (NIDA) (NIH); National Institute of Allergy and Infectious Diseases (NIAID) (NIH); NIH Office of AIDS Research (OAR) (NIH); National Institute of Mental Health (NIMH) (NIH); National Institute of Neurological Disorders and Stroke (NINDS) (NIH); National Institute on Deafness and Other Communication Disorders (NIDCD) (NIH); National Heart, Lung, and Blood Institute (NHLBI) (NIH); National Institute of Dental and Craniofacial Research (NIDCR) (NIH); National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH); Tulane University School of Medicine (Other)
Responsible Party: Principal Investigator, Paige Williams, Senior Lecturer on Biostatistics, Harvard School of Public Health (HSPH)
Other Study IDs: 1P01HD103133 - PH300; PH300 (Other: PHACS Protocol Number); 1P01HD103133 (NIH)
Record Dates: First submitted 2014-04-10; First posted 2014-04-22 (Estimated); Last update posted 2025-06-27 (Actual); Status verified 2025-06

CONDITIONS: HIV/AIDS
Keywords: HIV/AIDS, perinatal HIV infection
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Plasma, serum, peripheral blood mononuclear cells (PBMCs), urine, throat wash/gargle, saliva, and vaginal swabs.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Infected Cohort - Closed to accrual: Perinatally HIV-infected participants at or beyond their 18th birthday at enrollment.
- Uninfected Cohort: Perinatally HIV-exposed but uninfected participant at or beyond their 18th birthday at enrollment. May have horizontally-acquired HIV infection.

SUMMARY:
This is a prospective cohort study designed to define the impact of HIV infection and antiretroviral therapy (ART) on young adults with perinatal HIV infection (YAPHIV) as they transition into adulthood. A group of of perinatally exposed but uninfected young adults from a similar sociodemographic background and age distribution will be enrolled for comparison.

DETAILED DESCRIPTION:
AMP Up aims to define the impact of HIV infection and antiretroviral therapy (ART) on young adults with perinatal HIV infection as they transition into adulthood. A group of uninfected perinatally-exposed young adults from a similar sociodemographic background and age distribution will be enrolled for comparison.

The primary objectives of this study are:

* To identify infectious and non-infectious complications of HIV disease and toxicities resulting from long-term ART, including disease progression, immune dysfunction, viral resistance, end-organ disease, and mortality.
* To define the impact of HIV infection and ART on the long-term clinical outcomes of young adults, including:

  * Metabolic abnormalities and risk factors for cardiovascular disease, including glucose and lipid metabolism, blood pressure, and body composition.
  * Sexually transmitted infections (Chlamydia trachomatis, Neisseria gonorrhoeae, Trichomonas vaginalis, syphilis, human papillomavirus (HPV), genital warts and HSV) among males and females, and cervical HPV-associated pre-cancers and cancers and Mycoplasma genitalium and other vaginal microbiota among females.
  * Reproductive health, fertility, and pregnancy outcomes including mother-to-child transmission of HIV.
* To define the impact of perinatal HIV infection, its concomitant risk factors and ART on long-term neurocognitive and behavioral health outcomes, including:

  * Mental health and neurocognitive functioning.
  * Health care behaviors, including adherence to ART, participation in health care services, and transition to adult clinical care.
  * Risk behaviors, including sexual behavior and substance use.
  * Independent living skills, and vocational and education achievement necessary for successful transition to adult functioning and quality of life.

ELIGIBILITY:
Perinatally HIV-Infected Cohort

Inclusion Criteria:

* Perinatal HIV infection as documented in the medical record
* At or beyond their 18th birthday at the time of informed consent with no upper age limit
* Willing to provide access to existing medical records

  * Available medical record documentation since early childhood of:

    * ART exposure history
    * Opportunistic infection prophylaxis exposure history
    * Viral load and CD4+ cell count history
    * Major medical events history
* Willingness to participate and provide legal written consent

Exclusion Criteria:

* HIV acquired by other than maternal-child transmission (e.g., blood products, sexual contact, and IV drug use) as documented in the medical record

Uninfected Cohort

Inclusion Criteria:

* Absence of perinatal HIV infection as indicated in the medical record; the Perinatally HIV-Exposed Uninfected (PHEU) participant may have horizontally-acquired HIV infection
* At or beyond their 18th birthday at the time of informed consent with no upper age limit
* Willingness to participate and provide legal written consent

Exclusion Criteria:

* Have confirmed perinatal HIV infection as documented in the medical record

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Young adults 18 years of age or older at the time of enrollment with or without perinatal HIV-infection.
Sampling Method: Non-Probability Sample
Enrollment: 818 (Actual)
Dates: Start 2014-04 (Actual); Primary Completion 2025-05-31 (Actual); Study Completion 2025-05-31 (Actual)

PRIMARY OUTCOMES:
HIV disease progression | Annually for 6 years
  Factors of interest for this outcome include virologic suppression, immune impairment, immune activation, changes in ART, cumulative exposure to specific ART, viral resistance, co-infections, and host genetic polymorphisms. Data will be collected through chart abstraction and laboratory assessments and central laboratory testing.
Metabolic abnormalities | Annually for 6 years
  Factors of interest include BMI, body composition, systolic and diastolic blood pressure, lipid levels (total cholesterol, HDL cholesterol, LDL cholesterol, and triglycerides). Data will be collected by chart review, physical assessments, and laboratory evaluations.
Sexually transmitted infections (STI) | Annually for 6 years
  STI testing and chart review conducted annually.
Pregnancies | Annually for 6 years
  Data collected annually through online surveys and chart abstraction.
Mental health problems | Annually for 6 years
  Assessed at annually through the Patient Health Questionnaire (PHQ-9)) and General Anxiety Disorder-7 (GAD-7)
ART adherence | Annually for 6 years
  Data collected annually through an online survey.
Prevalence of risk behaviors including risky sexual behavior and licit and illicit substance use | Annually for 6 years
  Participants will complete an annual online survey.
Transition to adult functioning | Every 3 years for 6 years
  Every year participants will complete an online survey to collect data on educational attainment, employment, independent living and quality of life.
Hearing dysfunction | Every 3 years for 6 years
  Assessed through the NIH Toolbox and a questionnaire to be completed at Entry, Year 3 and Year 6 visits.
Language development | Once, at the Entry or Year 3 visit
  The Clinical Evaluation of Language Fundamentals (CELF) IV assessment will be completed at the Entry or Year 3 visit.
End-organ disease | Annually for 6 years
  Factors of interest for this outcome include virologic suppression, immune impairment, immune activation, changes in ART, cumulative exposure to specific ART, viral resistance, co-infections, and host genetic polymorphisms. Data will be collected through chart abstraction and laboratory assessments.
Mortality | Annually for 6 years
  Factors of interest for this outcome include virologic suppression, immune impairment, immune activation, changes in ART, cumulative exposure to specific ART, viral resistance, co-infections, and host genetic polymorphisms. Data will be collected through chart abstraction and laboratory assessments.
Risk factors for cardiovascular disease | Annually for 6 years
  Factors of interest include BMI, body composition, systolic and diastolic blood pressure, lipid levels (total cholesterol, HDL cholesterol, LDL cholesterol, and triglycerides) and cumulative cardiometabolic risk. Data will be collected by chart review, physical assessments, and laboratory evaluations.
Cervical HPV-associated pre-cancers and cancers (among female participants) | Annually for 6 years
  Data collected through annual chart review.
Cognitive impairment | Every 3 years for 6 years
  Assessed at Entry, Years 3, 6, 9, and 12 visits through the NIH Toolbox.
Maternal-to-child HIV transmission | Annually for 6 years
  Data collected through annual chart review.

CONTACTS AND LOCATIONS:
Overall Officials: Paige L Williams, Principal Investigator — Harvard School of Public Health (HSPH); Russell Van Dyke, MD, Principal Investigator — Tulane University School of Medicine; Katherine Tassiopoulos, DSc, MPH, Principal Investigator — Harvard School of Public Health (HSPH)
Locations (14):
- United States (13):
  - University of California San Diego, La Jolla, California
  - University of Colorado Denver Health Sciences Center, Aurora, Colorado
  - Children's Diagnostic and Treatment Center, Fort Lauderdale, Florida
  - University of Miami, Miami, Florida
  - Ann and Robert H. Lurie Children's Hospital, Chicago, Illinois
  - Tulane University Health Sciences Center, New Orleans, Louisiana
  - Children's Hospital Boston, Boston, Massachusetts
  - Rutgers - New Jersey Medical School, Newark, New Jersey
  - Bronx Lebanon Hospital Center, The Bronx, New York
  - Jacobi Medical Center, The Bronx, New York
  - St. Christopher's Hospital for Children, Philadelphia, Pennsylvania
  - St. Jude Children's Research Hospital, Memphis, Tennessee
  - Baylor College of Medicine, Houston, Texas
- San Juan Research Hospital, San Juan, Puerto Rico

REFERENCES:
- [Result] Tassiopoulos K, Patel K, Alperen J, Kacanek D, Ellis A, Berman C, Allison SM, Hazra R, Barr E, Cantos K, Siminski S, Massagli M, Bauermeister J, Siddiqui DQ, Puga A, Van Dyke R, Seage GR 3rd; Pediatric HIV/AIDS Cohort Study. Following young people with perinatal HIV infection from adolescence into adulthood: the protocol for PHACS AMP Up, a prospective cohort study. BMJ Open. 2016 Jun 9;6(6):e011396. doi: 10.1136/bmjopen-2016-011396. PMID 27288383
- [Result] Williams PL, Jesson J. Growth and pubertal development in HIV-infected adolescents. Curr Opin HIV AIDS. 2018 May;13(3):179-186. doi: 10.1097/COH.0000000000000450. PMID 29432228
- [Result] Innes S, Patel K. Noncommunicable diseases in adolescents with perinatally acquired HIV-1 infection in high-income and low-income settings. Curr Opin HIV AIDS. 2018 May;13(3):187-195. doi: 10.1097/COH.0000000000000458. PMID 29432231
- [Result] Goodenough CJ, Patel K, Van Dyke RB; Pediatric HIV/AIDS Cohort Study (PHACS). Is There a Higher Risk of Mother-to-child Transmission of HIV Among Pregnant Women With Perinatal HIV Infection? Pediatr Infect Dis J. 2018 Dec;37(12):1267-1270. doi: 10.1097/INF.0000000000002084. PMID 29742647
- [Result] Wilkinson JD, Williams PL, Yu W, Colan SD, Mendez A, Zachariah JPV, Van Dyke RB, Shearer WT, Margossian RE, Lipshultz SE; Pediatric HIV/AIDS Cohort Study (PHACS). Cardiac and inflammatory biomarkers in perinatally HIV-infected and HIV-exposed uninfected children. AIDS. 2018 Jun 19;32(10):1267-1277. doi: 10.1097/QAD.0000000000001810. PMID 29596110
- [Result] Alperen J, Davidson J, Siminski S, Seage GR 3rd; Pediatric HIV/AIDS Cohort Study. Utility of the National Death Index in Identifying Deaths in a Clinic-Based, Multisite Cohort: The Experience of the Pediatric HIV/AIDS Cohort Study. J Acquir Immune Defic Syndr. 2018 Sep 1;79(1):e37-e39. doi: 10.1097/QAI.0000000000001763. No abstract available. PMID 29847477
- [Result] Kacanek D, Huo Y, Malee K, Mellins CA, Smith R, Garvie PA, Tassiopoulos K, Lee S, Berman CA, Paul M, Puga A, Allison S; Pediatric HIV/AIDS Cohort Study. Nonadherence and unsuppressed viral load across adolescence among US youth with perinatally acquired HIV. AIDS. 2019 Oct 1;33(12):1923-1934. doi: 10.1097/QAD.0000000000002301. PMID 31274538
- [Result] Moscicki AB, Karalius B, Tassiopoulos K, Yao TJ, Jacobson DL, Patel K, Purswani M, Seage GR; Pediatric HIV/AIDS Cohort Study. Human Papillomavirus Antibody Levels and Quadrivalent Vaccine Clinical Effectiveness in Perinatally Human Immunodeficiency Virus-infected and Exposed, Uninfected Youth. Clin Infect Dis. 2019 Sep 13;69(7):1183-1191. doi: 10.1093/cid/ciy1040. PMID 30927547
- [Result] Yildirim C, Garvie PA, Chernoff M, Wilkins ML, Patton ED, Williams PL, Nichols SL; Memory and Executive Functioning Study of the Pediatric HIV/AIDS Cohort Study. The Role of Pharmacy Refill Measures in Assessing Adherence and Predicting HIV Disease Markers in Youth with Perinatally-Acquired HIV (PHIV). AIDS Behav. 2019 Aug;23(8):2109-2120. doi: 10.1007/s10461-019-02468-x. PMID 30929147
- [Result] Patel K, Seage GR 3rd, Burchett SK, Hazra R, Van Dyke RB; Pediatric HIV/AIDS Cohort Study. Disparities in HIV Viral Suppression Among Adolescents and Young Adults by Perinatal Infection. Am J Public Health. 2019 Jul;109(7):e9. doi: 10.2105/AJPH.2019.305108. No abstract available. PMID 31166735
- [Result] Smith R, Huo Y, Tassiopoulos K, Rutstein R, Kapetanovic S, Mellins C, Kacanek D, Malee K; Pediatric HIV/AIDS Cohort Study (PHACS). Mental Health Diagnoses, Symptoms, and Service Utilization in US Youth with Perinatal HIV Infection or HIV Exposure. AIDS Patient Care STDS. 2019 Jan;33(1):1-13. doi: 10.1089/apc.2018.0096. PMID 30601062
- [Result] Torre P 3rd, Russell JS, Smith R, Hoffman HJ, Lee S, Williams PL, Yao TJ; Pediatric HIV/AIDS Cohort Study (PHACS). Words-in-Noise Test Performance in Young Adults Perinatally HIV Infected and Exposed, Uninfected. Am J Audiol. 2020 Mar 5;29(1):68-78. doi: 10.1044/2019_AJA-19-00042. Epub 2020 Jan 31. PMID 32004075
- [Result] Patel K, Karalius B, Powis K, Kacanek D, Berman C, Moscicki AB, Paul M, Tassiopoulos K, Seage GR 3rd; HIV/AIDS Cohort Study (PHACS). Trends in post-partum viral load among women living with perinatal HIV infection in the USA: a prospective cohort study. Lancet HIV. 2020 Mar;7(3):e184-e192. doi: 10.1016/S2352-3018(19)30339-X. Epub 2019 Dec 20. PMID 31870676
- [Result] Tassiopoulos K, Huo Y, Patel K, Kacanek D, Allison S, Siminski S, Nichols SL, Mellins CA; Pediatric HIV/AIDS Cohort Study (PHACS). Healthcare Transition Outcomes Among Young Adults With Perinatally Acquired Human Immunodeficiency Virus Infection in the United States. Clin Infect Dis. 2020 Jun 24;71(1):133-141. doi: 10.1093/cid/ciz747. PMID 31584617
- [Result] Berman CA, Kacanek D, Nichamin M, Wilson D, Davtyan M, Salomon L, Patel K, Reznick M, Tassiopoulos K, Lee S, Bauermeister J, Paul M, Aldape T, Seage Iii GR. Using Social Media and Technology to Communicate in Pediatric HIV Research: Qualitative Study With Young Adults Living With or Exposed to Perinatal HIV. JMIR Pediatr Parent. 2020 Jun 23;3(1):e20712. doi: 10.2196/20712. PMID 32540839
- [Result] Cantos K, Franke MF, Tassiopoulos K, Williams PL, Moscicki AB, Seage GR 3rd; Pediatric HIV/AIDS Cohort Study. Inconsistent Sexual Behavior Reporting Among Youth Affected by Perinatal HIV Exposure in the United States. AIDS Behav. 2021 Oct;25(10):3398-3412. doi: 10.1007/s10461-021-03268-y. Epub 2021 Apr 24. PMID 33893876
- [Result] Sirois PA, Huo Y, Nozyce ML, Garvie PA, Harris LL, Malee K, McEvoy R, Mellins CA, Nichols SL, Smith R, Tassiopoulos K; Pediatric HIV/AIDS Cohort Study. Ageing with HIV: a longitudinal study of markers of resilience in young adults with perinatal exposure to HIV, with or without perinatally acquired HIV. J Int AIDS Soc. 2022 Sep;25 Suppl 4(Suppl 4):e25982. doi: 10.1002/jia2.25982. PMID 36176020
- [Result] Torre P 3rd, Zhang ZJ, Hoffman HJ, Frederick T, Purswani M, Williams PL, Yao TJ; Pediatric HIV/AIDS Cohort Study (PHACS). Auditory Function in the Pediatric HIV/AIDS Cohort Study Adolescent Master Protocol Up Young Adults: A Pilot Study. J Acquir Immune Defic Syndr. 2023 Apr 1;92(4):340-347. doi: 10.1097/QAI.0000000000003145. PMID 36729663
- [Result] Lemon TL, Tassiopoulos K, Tsai AC, Cantos K, Escudero D, Quinn MK, Kacanek D, Berman C, Salomon L, Nichols S, Chadwick EG, Seage GR 3rd, Williams PL; Pediatric HIV/AIDS Cohort Study (PHACS). Health Insurance Coverage, Clinical Outcomes, and Health-Related Quality of Life Among Youth Born to Women Living With HIV. J Acquir Immune Defic Syndr. 2023 Jan 1;92(1):6-16. doi: 10.1097/QAI.0000000000003100. PMID 36150048
- [Result] Tassiopoulos K, Huo Y, Kacanek D, Malee K, Nichols S, Mellins CA, Kohlhoff S, Van Dyke RB; Pediatric HIV/AIDS Cohort Study. Association of Perceived Social Support with Viral Suppression Among Young Adults with Perinatally-Acquired HIV in the US-based Pediatric HIV/AIDS Cohort Study (PHACS). Clin Epidemiol. 2023 May 9;15:601-611. doi: 10.2147/CLEP.S403570. eCollection 2023. PMID 37193342
- [Result] Dirajlal-Fargo S, Yu W, Jacobson DL, Mirza A, Geffner ME, Jao J, McComsey GA; Pediatric HIV/AIDS Cohort Study (PHACS). Gut permeability is associated with lower insulin sensitivity in youth with perinatally acquired HIV. AIDS. 2024 Jul 1;38(8):1163-1171. doi: 10.1097/QAD.0000000000003896. Epub 2024 Mar 28. PMID 38564437
- [Result] Gojanovich GS, Yu W, Zhang ZJ, Jacobson DL, Yao TJ, Jao J, Libutti DE, Geffner ME, Gerschenson M; Pediatric HIV/AIDS Cohort Study. Longitudinal changes in mitochondrial-associated measures and insulin resistance in youth with perinatally-acquired HIV in the U.S. Mitochondrion. 2024 Sep;78:101936. doi: 10.1016/j.mito.2024.101936. Epub 2024 Jul 14. PMID 39009104
- See also: Pediatric HIV/AIDS Cohort Study — http://www.phacsstudy.org